CLINICAL TRIAL: NCT03844542
Title: Therapeutic Plasma Exchange in the Treatment of Sepsis Associated Multi-Organ Failure [SAMOF-TPE]
Acronym: SAMOF-TPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Forsyth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1187
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Plasma Exchange

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Therapeutic plasma exchange (Experimental): Perform therapeutic plasma exchange in addition to standard care for patients with sepsis induced multi-organ failure
  Interventions: Device: Therapeutic plasma exchange
- Standard care alone for sepsis (No Intervention): Standard care for patients with sepsis induced multi-organ failure

INTERVENTIONS:
Device: Therapeutic plasma exchange — Perform therapeutic plasma exchange in patients with sepsis induced multi-organ failure
  Arms: Therapeutic plasma exchange

SUMMARY:
The investigators prospective, randomized adult clinical trial investigates the therapeutic efficacy of early therapeutic plasma exchange as adjunct treatment to standard therapy in patients with refractory septic shock and multiple organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients are eligible for inclusion if they have sepsis with refractory shock and evidence of organ failure.

Exclusion Criteria:

* Persons who are pregnant
* Persons who are incarcerated
* Acute surgical catastrophe without potential for intervention or source control
* Cardiac arrest with unknown neurologic status, including patients being treated with therapeutic hypothermia
* Presence of severe acute brain injury or severe dementia
* Cardiogenic, neurogenic, obstructive, or post-cardiotomy shock
* Acute pancreatitis with no established source of infection
* Diabetic ketoacidosis as primary pathology

  * Note: Septic patients who develop DKA are eligible for inclusion. However, patients in whom organ dysfunction and hemodynamic instability are due primarily to volume depletion and acidosis from DKA should not be included.
* Need for mechanical circulatory support
* Prolonged acute illness with > 24 hours of pressor needs at enrollment and/or end organ damage with further care deemed to be "futile."

  * NOTE: The time resets if a new inciting event leads to SAMOF.
  * For example, if a patient has sepsis stabilized but requires operative intervention for source control within the initial 24 hours of admission and returns to the ICU with SAMOF, the patient is again eligible for randomization for the next 24 hours.
* Bedbound state or poor baseline functional status with ECOG performance status score ≥ 3
* Underlying terminal illness/malignancy with < 6 months life expectancy
* Advanced chronic liver disease/cirrhosis with evidence of portal hypertension
* Asplenia
* HIV with HARRT non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
28-Day Mortality | 28 days
  28 days

IPD SHARING:
Plan to Share IPD: Undecided